CLINICAL TRIAL: NCT04765709
Title: BRIDGE Trial: Phase II Trial of durvalumaB and chemotheRapy Induction Followed by Durvalumab and Radiotherapy in larGe volumE Stage III NSCLC
Brief Title: Durvalumab and Chemotherapy Induction Followed by Durvalumab and Radiotherapy in Large Volume Stage III NSCLC
Acronym: BRIDGE
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low enrolment rate
Sponsor: Mario Negri Institute for Pharmacological Research (Other)
Collaborators: AstraZeneca (Industry); Fondazione IRCCS Istituto Nazionale dei Tumori, Milano (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRFMN-NSCLC-8187; 2019-004025-24 (EudraCT Number)
Record Dates: First submitted 2021-02-08; First posted 2021-02-21 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-03

CONDITIONS: Non-small Cell Lung Cancer Stage III
Keywords: Carcinoma, Non-Small-Cell Lung; Radiotherapy; Immunotherapy; durvalumab; Stage III; Unresectable NSCLC; Phase II; Concomitant immuno-radiotherapy; Concomitant immuno-chemotherapy; Chemotherapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — durvalumab; Platinum Compounds; Cisplatin; Carboplatin; Vinorelbine; Pemetrexed; Radiotherapy

STUDY DESIGN:
Intervention Model Description: multicentric, open label, single arm, minimax Simon 2 stages, phase 2 trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- BRIDGE single arm (Experimental): Treatment plan:
  * Part 1: induction with durvalumab plus histology-based chemotherapy regimen.
  * Part 2: patients with a sufficient tumor shrinkage to be considered eligible for part 2 and they will be treated concomitantly with durvalumab and radiotherapy.
  * Part 3: patients with partial response or stable disease after part 2 will be eligible for durvalumab maintenance, for up to 2 years or until disease progression or unacceptable toxicity.
  Interventions: Combination Product: durvalumab plus platinum-based chemotherapy (cisplatin or carboplatin plus vinorelbine or pemetrexed); Combination Product: Durvalumab plus radiotherapy; Biological: durvalumab

INTERVENTIONS:
Combination Product: durvalumab plus platinum-based chemotherapy (cisplatin or carboplatin plus vinorelbine or pemetrexed) — Induction therapy: durvalumab plus histology-based chemotherapy regimen (cisplatin or carboplatin plus vinorelbine for squamous histology and pemetrexed for non-squamous histology).
Combination Product: Durvalumab plus radiotherapy — Concomitant durvalumab and radiotherapy
Biological: durvalumab — Consolidation treatment with durvalumab

SUMMARY:
Standard treatment for stage III Non-Small Cells Lung Cancer (NSCLC) not eligibile for surgery is concomitant chemoradiotherapy. However median progression free survival and overall survival is still poor with only 15% of patients alive at 5 years. The addition of maintenance therapy with durvalumab after chemoradiation showed a significant benefit in PFS and OS, with good tolerability and no concerns in terms of safety. However, about 30% of patients with stage III are not eligible to concurrent chemoradiotherapy because of large volumes of the tumor. To date, these patients are initially treated with chemotherapy with the aim of reducing tumor volumes and allowing sequential radiotherapy. Response rate ranges between 25-30% and majority of patients will not become suitable for radiotherapy.

The combination of immunotherapy plus standard chemotherapy in advanced stages doubles response rates and provides major tumor shrinkage compared to standard chemotherapy alone. For these reasons, the investigators want to exploit the synergistic effect of immunotherapy combined with chemotherapy in the induction phase, in order to render suitable for radiotherapy a larger number of patients, and in a second phase the synergistic effect with radiotherapy.

Based on these premises the investigators designed a single arm, phase 2 trial to determine the efficacy and safety of combining immunotherapy with the drug durvalumab in association with standard chemotherapy and subsequently with standard radiotherapy, followed by a treatment of maintenance with only durvalumab.

The study population includes patients with NSCLC not eligible for surgery or concurrent chemoradiation at diagnosis because of large tumor volumes.

BRIDGE trial aims to evaluate the proportion of patients who did not progress and who achieved a mean lung dose <20 Gy and/or a lung V20<35% (response) after part 1. The primary objective of the study is to increase the proportion of patients eligible for immunotherapy plus radiotherapy after induction with durvalumab and chemotherapy, in comparison with historical controls.

This study will last approximately 60 months and will include approximately 65 eligible patients in 3 international cancer centres of excellence.

DETAILED DESCRIPTION:
Standard treatment for stage III Non-Small Cells Lung Cancer (NSCLC) not eligibile for surgery is concomitant chemoradiotherapy. However median progression free survival and overall survival is still poor with only 15% of patients alive at 5 years. The addition of maintenance therapy with durvalumab after chemoradiation showed a significant benefit in PFS and OS, with good tolerability and no concerns in terms of safety. However, about 30% of patients with stage III are not eligible to concurrent chemoradiotherapy because of large volumes of the tumor. To date, these patients are initially treated with chemotherapy with the aim of reducing tumor volumes and allowing sequential radiotherapy. Response rate ranges between 25-30% and majority of patients will not become suitable for radiotherapy.

The combination of immunotherapy plus standard chemotherapy in advanced stages doubles response rates and provides major tumor shrinkage compared to standard chemotherapy alone. For these reasons, the investigators want to exploit the synergistic effect of immunotherapy combined with chemotherapy in the induction phase, in order to render suitable for radiotherapy a larger number of patients, and in a second phase the synergistic effect with radiotherapy.

Based on these premises the investigators designed a single arm, phase 2 trial to determine the efficacy and safety of combining immunotherapy with the drug durvalumab in association with standard chemotherapy and subsequently with standard radiotherapy, followed by a treatment of maintenance with only durvalumab.

The study population includes patients with NSCLC not eligible for surgery or concurrent chemoradiation at diagnosis because of large tumor volumes.

The study consists of 3 parts:

* Part 1: induction with durvalumab plus chemotherapy.
* Part 2: patients with a sufficient tumor shrinkage to be considered eligible for part 2 and they will be treated concomitantly with durvalumab and radiotherapy.
* Part 3: patients with partial response or stable disease after part 2 will be eligible for durvalumab maintenance, for up to 2 years or until disease progression or unacceptable toxicity.

BRIDGE trial aims to evaluate the proportion of patients who did not progress and who achieved a mean lung dose <20 Gy and/or a lung V20<35% (response) after part 1. The primary objective of the study is to increase the proportion of patients eligible for immunotherapy plus radiotherapy after induction with durvalumab and chemotherapy, in comparison with historical controls.

This study will last approximately 60 months and will include approximately 65 eligible patients in 3 international cancer centres of excellence.

ELIGIBILITY:
Inclusion Criteria

FOR PART 1 (INDUCTION CHEMOTHERAPY IN ASSOCIATION WITH DURVALUMAB):

1. Capable of giving signed informed consentwhich includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol. Written informed consent and any locally required authorization (eg, European Union [EU] Data Privacy Directive in the EU) obtained from the patient/legal representative prior to performing any protocol-related procedures, including screening evaluations.
2. Age > 18 years at time of study entry
3. Histologically- or cytologically-documented NSCLC, in locally advanced (Stage III-v.8 IASLC)
4. Eligible for platinum-based chemotherapy (platinum - pemetrexed for non-squamous and platinum-vinorelbine for squamous histology)
5. Patients not eligible for surgery and chemoradiation for Dosimetry not meeting the following constraints to organs at risk (Kong 2011, Marks 2010, De Ruysscher 2017, Marks 2010, Gagliardi 2010, Wang 2017, Antonia 2017, Kirkpatrick 2010):

   * Total mean lung dose (Right Lung+Left Lung-GTV) < 20 Gy and/or
   * Lung V20 defined as percentage of normal parenchyma receiving 20 Gy or more (Right Lung+Left Lung-PTV) < 35%
   * Heart V45 <30% and/or Mean Heart Dose <20 Gy

   If the dosimetry criteria are met, other clinical conditions for avoiding concurrent chemoradiation are:
   * Bilateral supraclavicular involvement
   * Contralateral mediastinal and/or hilar involvement
   * Primary tumor > 7 cm or several nodules in different lobes of the same lung or bulky mediastinal lymphonodes.

   Each patient will be discussed in a web multidisciplinary team among all the three involved Cancer Core Europe [CCE] centers. If dosimetry criteria are met, patient not eligible for surgery and chemoradiation due to other clinical condition(s) will be specifically defined and confirmed by at least 2 out of 3 CCE
6. Tumor sample requirements: availability of an archived tumour tissue block (or unstained slides to perform local PDL1 assessment following protocol procedure)
7. Patient's willingness to undergo blood draws to provide plasma and blood samples for analysis according to study objectives
8. Patients without history of previous radiotherapy. Patients with previous radiotherapy performed to the thorax, including radiotherapy for breast cancer, especially in the last 10 years, have to be discussed case by case in the Multidisciplinary Team Meeting
9. Life expectancy ≥12 weeks at the start of treatment
10. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
11. Evidence of post-menopausal status or negative urinary or serum pregnancy test for female pre-menopausal patients. Women will be considered post-menopausal if they have been amenorrheic for 12 months without an alternative medical cause. The following age-specific requirements apply:

    1. Women <50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of exogenous hormonal treatments and if they have luteinizing hormone and follicle- stimulating hormone levels in the post-menopausal range for the institution or underwent surgical sterilization (bilateral oophorectomy or hysterectomy).
    2. Women ≥50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of all exogenous hormonal treatments, had radiation-induced menopause with last menses >1 year ago, had chemotherapy-induced menopause with last menses >1 year ago, or underwent surgical sterilization (bilateral oophorectomy, bilateral salpingectomy or hysterectomy).
12. Patient willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up.
13. Adequate normal organ and marrow function as defined below:

    * Haemoglobin ≥9.0 g/dL (5.59 mmol/L)
    * Absolute neutrophil count (ANC) > 1.5 x 109/L (> 1500/mm3)
    * Platelet count ≥100 x 109/L (100000/mm3)
    * Serum bilirubin ≤1.5 x institutional upper limit of normal (ULN). This will not apply to patients with confirmed Gilbert's syndrome (persistent or recurrent hyperbilirubinemia that is predominantly unconjugated in the absence of hemolysis or hepatic pathology), who will be allowed only in consultation with their physician.
    * AST (SGOT)/ALT (SGPT) ≤2.5 x institutional upper limit of normal
    * Adequate renal function defined as normal serum creatinine levels or calculated creatinine clearance (according to Cockroft-Gault or by 24 hour-urine collection): ≥60 ml/min for patient receiving cisplatin ≥45 ml/min for patient receiving carboplatin.
14. Body weight > 30 Kg
15. Absence of a known severe hypersensitivity (≥ Grade 3) to any of the study chemotherapy agents and/or to durvalumab and/or to any of their excipients.

FOR PART 2 (RADIOTHERAPY CONCURRENTLY WITH DURVALUMAB):

1. Absence of progressive disease by RECIST 1.1 together with evidence of tumor shrinkage at the evaluation conducted at the end of part 1. Whether the degree of tumor shrinkage will be sufficient to consider the patient eligible for part 2 will be discussed in a web multidisciplinary team among involved CCE centers.
2. ECOG Performance Status of 0 - 1
3. Absence of dyspnea of minimal exertion or oxygen requirement after CT+D
4. Sufficient PFTs performed after the last cycle of CT+D:

   * FEV1 > 1L or ≥ 30%
   * DLCO > 30%
5. The patient's dosimetry must meet the following constraints to organs at risk (Kong 2011, Marks 2010, De Ruysscher 2017, Marks 2010, Gagliardi 2010, Wang 2017, Antonia 2017, Kirkpatrick 2010):

   * Spinal cord maximum dose < 50 Gy
   * Total mean lung dose (Right Lung+Left Lung-GTV) < 20 Gyand/or
   * Lung V20 defined as percentage of normal parenchyma receiving 20 Gy or more (Right Lung+Left Lung-PTV) < 35%
   * Heart V45 <30% and/or Mean Heart Dose <20 Gy
6. In case of dosimetry criteria met before part 1, confirmed resolution of clinical condition(s) that led to initial inegibility. The resolution of the clinical condition is discussed in the multidisciplinary team, at least 2 out of 3 CCE must agree.

FOR PART 3 (MAINTENANCE WITH DURVALUMAB):

1. Evidence of partial response or stable disease at the evaluation conducted at the end of Part 2
2. Absence of grade 2-3 pneumonitis

Exclusion Criteria:

1. Stage IV NSCLC
2. Patient amenable to curative intent surgery or concurrent chemoradiation
3. Mixed small cell and non-small cell lung cancer histology
4. Patients who already received therapy for locally advanced NSCLC
5. Dyspnea of minimal exertion or oxygen requirement
6. Recent medical history of cardiac events during the last 6 months (ischemic or congestive heart failure)
7. Pancoast tumors
8. Prior exposure to any anti-PD-1 or anti-PD-L1 antibody, including durvalumab
9. Participation in another clinical study with an investigational product during the last 4 weeks, unless it is an observational (non-interventional) clinical study or during the follow-up period of an interventional study
10. Any concurrent chemotherapy, immunotherapy, biologic, or hormonal therapy for cancer treatment. Concurrent use of hormonal therapy for non-cancer-related conditions (e.g., hormone replacement therapy) is acceptable.
11. Active or prior documented autoimmune disease within the past 2 years or inflammatory disorders (including inflammatory bowel disease [e.g., colitis or Crohn's disease], diverticulitis [with the exception of diverticulosis], systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc]). The following are exceptions to this criterion:

    1. Patients with vitiligo or alopecia
    2. Patients with Grave's disease not requiring systemic treatment within the past 2 years
    3. Patients with hypothyroidism (e.g., following Hashimoto syndrome) stable on hormone replacement
    4. Any chronic skin condition that does not require systemic therapy (e.g. patients with psoriasis not requiring systemic treatment within the past 2 years)
    5. Patients without active disease in the last 2 years may be included but only after consultation with the study physician
    6. Patients with celiac disease controlled by diet alone
12. Uncontrolled intercurrent illness including, but not limited to, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, active peptic ulcer disease or gastritis, active bleeding diatheses, ongoing or active infection, including any patient known to have evidence of acute or chronic hepatitis B (positive HBV surface antigen (HBsAg) result), hepatitis C, human immunodeficiency virus (HIV) (positive HIV 1/2 antibodies) or tuberculosis (clinical evaluation that includes clinical history, physical examination and radiographic findings, and TB testing in line with local practice), psychiatric illness/social situations that would limit compliance with study requirements or compromise the ability of the patient to give written informed consent. [Patients with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody [anti-HBc] and absence of HBsAg) are eligible. Patients positive for hepatitis C (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA.]
13. History of another primary malignancy except for

    1. Malignancy treated with curative intent and with no known active disease ≥3 years before the first dose of study drug and of low potential risk for recurrence
    2. Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease
    3. Adequately treated carcinoma in situ without evidence of disease, e.g. cervical cancer in situ
    4. Superficial bladder cancer without evidence of disease
14. Female patients who are pregnant or breastfeeding or male or female patients of reproductive potential who are not willing to employ effective birth control from screening to 90 days after the last dose of durvalumab monotherapy
15. Any unresolved toxicity NCI CTCAE Grade ≥2 from previous anticancer therapy with the exception of alopecia, vitiligo, and the laboratory values defined in the inclusion criteria

    1. Patients with Grade ≥2 neuropathy will be evaluated on a case-by-case basis after consultation with the Study Physician.
    2. Patients with irreversible toxicity not reasonably expected to be exacerbated by treatment with durvalumab may be included only after consultation with the Study Physician.
16. Major surgical procedure (as defined by the Investigator) within 28 days prior to the first dose of investigational product.
17. History of allogenic organ transplantation.
18. Mean QT interval corrected for heart rate using Fridericia's formula (QTcF) ≥470 ms
19. History of active primary immunodeficiency
20. Current or prior use of immunosuppressive medication within 14 days before the first dose of durvalumab. The following are exceptions to this criterion:

    1. Intranasal, inhaled, topical steroids, or local steroid injections (e.g., intra articular injection)
    2. Systemic corticosteroids at physiologic doses not to exceed 10 mg daily of prednisone or its equivalent
    3. Steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication) Systemic steroid administration required as prophylaxis against or to manage toxicities arising from chemotherapy and/or radiotherapy delivered as part of therapy for locally advanced NSCLC is allowed
21. Receipt of live attenuated vaccine within 30 days prior to the first dose of IP. Note: Patients, if enrolled, should not receive live vaccine whilst receiving IP and up to 30 days after the last dose of IP.
22. Known allergy or hypersensitivity to any of the study drugs or any of the study drug excipients.
23. Judgment by the investigator that the patient is unsuitable to participate in the study and the patient is unlikely to comply with study procedures, restrictions and requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-09-24 (Actual); Primary Completion 2025-01-30 (Actual); Study Completion 2025-01-30 (Actual)

PRIMARY OUTCOMES:
Proportion of patients who did not progressed and who achieved a mean lung dose <20 Gy and/or a lung V20<35% (response) after part 1 | At the end of part 1 of induction chemo-immunotherapy/before part 2 (assessed up to 60 months)
  The primary objective of the study is to increase the proportion of patients eligible for immunotherapy plus radiotherapy after induction with durvalumab and chemotherapy, in comparison to historical controls.

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) of patients receiving durvalumab and chemotherapy induction followed by immuno-radiotherapy and durvalumab consolidation. | From the date of start of induction chemo-immunotherapy until the date of first documented progression or death from any cause, whichever came first (assessed up to 60 months)
  PFS is defined as the time from the date of start of induction treatment until the date of objective disease progression or death to any cause whichever comes first. PFS will be evaluated using RECIST 1.1 criteria according to investigators and blinded central review (BCR).
Proportion of patients with complete response or partial response (as best response) | Assessed up to 60 months
  To evaluate Objective Response Rate (ORR) of each phase of treatment and the overall response rate. ORR is defined as the proportion of patients with complete or partial response (as best response) according to RECIST 1.1 as assessed by Investigators and BCR.
Overall Survival (OS) of patients receiving durvalumab and chemotherapy induction followed by immuno-radiotherapy and durvalumab consolidation. | Assessed up to 60 months
  OS is defined as the time from the date of start of induction treatment until death due to any cause. Patients alive at the time of statistical analysis will be censored at their last information on vital status.
Frequency and nature of adverse reactions (ARs) and Serious Adverse Events (SAEs) (toxicity and safety). | Assessed up to 60 months
  The assessment of safety will be mainly based on adverse reactions (ARs) and the frequency and nature of SAEs. Toxicity and safety will be evaluated during each part of the program, throughout study duration.

OTHER OUTCOMES:
Concordance between patients who reach the primary endpoint and patients who are included in part 2 after the evaluation of the multidisciplinary team | Assessed up to 60 months
  To evaluate the concordance between patients who reach the primary endpoint and patients who are included in part 2 after the evaluation of the multidisciplinary team
PD-L1 expression as predictive biomarker for clinical outcomes | Assessed up to 60 months
  To evaluate correlation of clinical outcome with PD-L1 expression (in percentage %).
Dynamic changes in mutations in coding area of Cell-Free DNA (cfDNA) in correlation with response | Assessed up to 60 months
  Plasma for cfDNA will be analyzed through whole exome sequencing (considering coding region only) to assess correlation with response.
Dynamic changes in mutations in coding area of a tumor genome (on Blood-based Tumor Mutational Burden, bTMB) | Assessed up to 60 months
  To assess the dynamic changes of the tumor mutational profile upon different treatment time points.

CONTACTS AND LOCATIONS:
Overall Officials: Valter Torri, Study Chair — Istituto Di Ricerche Farmacologiche Mario Negri; Roberto Ferrara, Principal Investigator — Fondazione IRCCS ISTITUTO NAZIONALE TUMORI
Locations (3):
- Gustave Roussy Institute, Paris, France
- Fondazione IRCCS Istituto Nazionale dei Tumori, Milan, Italy
- Vall d'Hebron Barcelona Hospital, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alexandrov LB, Nik-Zainal S, Wedge DC, Aparicio SA, Behjati S, Biankin AV, Bignell GR, Bolli N, Borg A, Borresen-Dale AL, Boyault S, Burkhardt B, Butler AP, Caldas C, Davies HR, Desmedt C, Eils R, Eyfjord JE, Foekens JA, Greaves M, Hosoda F, Hutter B, Ilicic T, Imbeaud S, Imielinski M, Jager N, Jones DT, Jones D, Knappskog S, Kool M, Lakhani SR, Lopez-Otin C, Martin S, Munshi NC, Nakamura H, Northcott PA, Pajic M, Papaemmanuil E, Paradiso A, Pearson JV, Puente XS, Raine K, Ramakrishna M, Richardson AL, Richter J, Rosenstiel P, Schlesner M, Schumacher TN, Span PN, Teague JW, Totoki Y, Tutt AN, Valdes-Mas R, van Buuren MM, van 't Veer L, Vincent-Salomon A, Waddell N, Yates LR; Australian Pancreatic Cancer Genome Initiative; ICGC Breast Cancer Consortium; ICGC MMML-Seq Consortium; ICGC PedBrain; Zucman-Rossi J, Futreal PA, McDermott U, Lichter P, Meyerson M, Grimmond SM, Siebert R, Campo E, Shibata T, Pfister SM, Campbell PJ, Stratton MR. Signatures of mutational processes in human cancer. Nature. 2013 Aug 22;500(7463):415-21. doi: 10.1038/nature12477. Epub 2013 Aug 14. PMID 23945592
- [Background] Antonia SJ, Villegas A, Daniel D, Vicente D, Murakami S, Hui R, Yokoi T, Chiappori A, Lee KH, de Wit M, Cho BC, Bourhaba M, Quantin X, Tokito T, Mekhail T, Planchard D, Kim YC, Karapetis CS, Hiret S, Ostoros G, Kubota K, Gray JE, Paz-Ares L, de Castro Carpeno J, Wadsworth C, Melillo G, Jiang H, Huang Y, Dennis PA, Ozguroglu M; PACIFIC Investigators. Durvalumab after Chemoradiotherapy in Stage III Non-Small-Cell Lung Cancer. N Engl J Med. 2017 Nov 16;377(20):1919-1929. doi: 10.1056/NEJMoa1709937. Epub 2017 Sep 8. PMID 28885881
- [Background] Antonia SJ, Villegas A, Daniel D, Vicente D, Murakami S, Hui R, Kurata T, Chiappori A, Lee KH, de Wit M, Cho BC, Bourhaba M, Quantin X, Tokito T, Mekhail T, Planchard D, Kim YC, Karapetis CS, Hiret S, Ostoros G, Kubota K, Gray JE, Paz-Ares L, de Castro Carpeno J, Faivre-Finn C, Reck M, Vansteenkiste J, Spigel DR, Wadsworth C, Melillo G, Taboada M, Dennis PA, Ozguroglu M; PACIFIC Investigators. Overall Survival with Durvalumab after Chemoradiotherapy in Stage III NSCLC. N Engl J Med. 2018 Dec 13;379(24):2342-2350. doi: 10.1056/NEJMoa1809697. Epub 2018 Sep 25. PMID 30280658
- [Background] Auperin A, Le Pechoux C, Rolland E, Curran WJ, Furuse K, Fournel P, Belderbos J, Clamon G, Ulutin HC, Paulus R, Yamanaka T, Bozonnat MC, Uitterhoeve A, Wang X, Stewart L, Arriagada R, Burdett S, Pignon JP. Meta-analysis of concomitant versus sequential radiochemotherapy in locally advanced non-small-cell lung cancer. J Clin Oncol. 2010 May 1;28(13):2181-90. doi: 10.1200/JCO.2009.26.2543. Epub 2010 Mar 29. PMID 20351327
- [Background] Bayman N, Blackhall F, McCloskey P, Taylor P, Faivre-Finn C. How can we optimise concurrent chemoradiotherapy for inoperable stage III non-small cell lung cancer? Lung Cancer. 2014 Feb;83(2):117-25. doi: 10.1016/j.lungcan.2013.11.017. Epub 2013 Dec 1. PMID 24373738
- [Background] Bracci L, Schiavoni G, Sistigu A, Belardelli F. Immune-based mechanisms of cytotoxic chemotherapy: implications for the design of novel and rationale-based combined treatments against cancer. Cell Death Differ. 2014 Jan;21(1):15-25. doi: 10.1038/cdd.2013.67. Epub 2013 Jun 21. PMID 23787994
- [Background] Bradley JD, Paulus R, Komaki R, Masters G, Blumenschein G, Schild S, Bogart J, Hu C, Forster K, Magliocco A, Kavadi V, Garces YI, Narayan S, Iyengar P, Robinson C, Wynn RB, Koprowski C, Meng J, Beitler J, Gaur R, Curran W Jr, Choy H. Standard-dose versus high-dose conformal radiotherapy with concurrent and consolidation carboplatin plus paclitaxel with or without cetuximab for patients with stage IIIA or IIIB non-small-cell lung cancer (RTOG 0617): a randomised, two-by-two factorial phase 3 study. Lancet Oncol. 2015 Feb;16(2):187-99. doi: 10.1016/S1470-2045(14)71207-0. Epub 2015 Jan 16. PMID 25601342
- [Background] Brahmer JR, Tykodi SS, Chow LQ, Hwu WJ, Topalian SL, Hwu P, Drake CG, Camacho LH, Kauh J, Odunsi K, Pitot HC, Hamid O, Bhatia S, Martins R, Eaton K, Chen S, Salay TM, Alaparthy S, Grosso JF, Korman AJ, Parker SM, Agrawal S, Goldberg SM, Pardoll DM, Gupta A, Wigginton JM. Safety and activity of anti-PD-L1 antibody in patients with advanced cancer. N Engl J Med. 2012 Jun 28;366(26):2455-65. doi: 10.1056/NEJMoa1200694. Epub 2012 Jun 2. PMID 22658128
- [Background] Brahmer JR, Horn L, Gandhi L, Spigel DR, Antonia SJ, Rizvi NA, et al. Nivolumab (anti-PD-1, BMS-936558, ONO-4538) in patients (pts) with advanced non-small-cell lung cancer (NSCLC): Survival and clinical activity by subgroup analysis [ASCO abstract 8112]. J Clin Oncol 2014;32(Suppl)
- [Background] Brookmeyer R, Crowley J. A confidence interval for the median survival time. Biometrics 1982, 38, 29-41. doi:10.2307/2530286
- [Background] Butte MJ, Keir ME, Phamduy TB, Sharpe AH, Freeman GJ. Programmed death-1 ligand 1 interacts specifically with the B7-1 costimulatory molecule to inhibit T cell responses. Immunity. 2007 Jul;27(1):111-22. doi: 10.1016/j.immuni.2007.05.016. Epub 2007 Jul 12. PMID 17629517
- [Background] De Ruysscher D, Reynders K, Van Limbergen E, Lambrecht M. Radiotherapy in combination with immune checkpoint inhibitors. Curr Opin Oncol. 2017 Mar;29(2):105-111. doi: 10.1097/CCO.0000000000000352. PMID 28085679
- [Background] De Ruysscher D, Faivre-Finn C, Moeller D, Nestle U, Hurkmans CW, Le Pechoux C, Belderbos J, Guckenberger M, Senan S; Lung Group and the Radiation Oncology Group of the European Organization for Research and Treatment of Cancer (EORTC). European Organization for Research and Treatment of Cancer (EORTC) recommendations for planning and delivery of high-dose, high precision radiotherapy for lung cancer. Radiother Oncol. 2017 Jul;124(1):1-10. doi: 10.1016/j.radonc.2017.06.003. Epub 2017 Jun 27. PMID 28666551
- [Background] Drake CG, McDermott DF, Sznol M, Choueiri TK, Kluger HM, Powderly JD et al. Survival, safety, and response duration results of nivolumab (Anti-PD-1; BMS-936558; ONO-4538) in a phase I trial in patients with previously treated metastatic renal cell carcinoma (mRCC): Long-term patient follow-up [abstract 4514]. J Clin Oncol 2013;31(Suppl)
- [Background] Dunn GP, Old LJ, Schreiber RD. The three Es of cancer immunoediting. Annu Rev Immunol. 2004;22:329-60. doi: 10.1146/annurev.immunol.22.012703.104803. PMID 15032581
- [Background] Eisenhauer EA, Therasse P, Bogaerts J, Schwartz LH, Sargent D, Ford R, Dancey J, Arbuck S, Gwyther S, Mooney M, Rubinstein L, Shankar L, Dodd L, Kaplan R, Lacombe D, Verweij J. New response evaluation criteria in solid tumours: revised RECIST guideline (version 1.1). Eur J Cancer. 2009 Jan;45(2):228-47. doi: 10.1016/j.ejca.2008.10.026. PMID 19097774
- [Background] Ellis S, Carroll KJ, Pemberton K. Analysis of duration of response in oncology trials. Contemp Clin Trials. 2008 Jul;29(4):456-65. doi: 10.1016/j.cct.2007.10.008. Epub 2007 Nov 12. PMID 18187370
- [Background] Fairman D, Narwal R, Liang M, Robbins PB, Schneider A, Chavez C, et al. Pharmacokinetics of durvalumab, a fully human anti-PDL1 monoclonal antibody, in patients with advanced solid tumours. Journal of Clinical Oncology, 2014 ASCO Annual Meeting Abstracts;32(5s): (suppl; abstr 2602)
- [Background] Fife BT, Bluestone JA. Control of peripheral T-cell tolerance and autoimmunity via the CTLA-4 and PD-1 pathways. Immunol Rev. 2008 Aug;224:166-82. doi: 10.1111/j.1600-065X.2008.00662.x. PMID 18759926
- [Background] Forde PM, Chaft JE, Smith KN, Anagnostou V, Cottrell TR, Hellmann MD, Zahurak M, Yang SC, Jones DR, Broderick S, Battafarano RJ, Velez MJ, Rekhtman N, Olah Z, Naidoo J, Marrone KA, Verde F, Guo H, Zhang J, Caushi JX, Chan HY, Sidhom JW, Scharpf RB, White J, Gabrielson E, Wang H, Rosner GL, Rusch V, Wolchok JD, Merghoub T, Taube JM, Velculescu VE, Topalian SL, Brahmer JR, Pardoll DM. Neoadjuvant PD-1 Blockade in Resectable Lung Cancer. N Engl J Med. 2018 May 24;378(21):1976-1986. doi: 10.1056/NEJMoa1716078. Epub 2018 Apr 16. PMID 29658848
- [Background] Gagliardi G, Constine LS, Moiseenko V, Correa C, Pierce LJ, Allen AM, Marks LB. Radiation dose-volume effects in the heart. Int J Radiat Oncol Biol Phys. 2010 Mar 1;76(3 Suppl):S77-85. doi: 10.1016/j.ijrobp.2009.04.093. PMID 20171522
- [Background] Gandhi L, Rodriguez-Abreu D, Gadgeel S, Esteban E, Felip E, De Angelis F, Domine M, Clingan P, Hochmair MJ, Powell SF, Cheng SY, Bischoff HG, Peled N, Grossi F, Jennens RR, Reck M, Hui R, Garon EB, Boyer M, Rubio-Viqueira B, Novello S, Kurata T, Gray JE, Vida J, Wei Z, Yang J, Raftopoulos H, Pietanza MC, Garassino MC; KEYNOTE-189 Investigators. Pembrolizumab plus Chemotherapy in Metastatic Non-Small-Cell Lung Cancer. N Engl J Med. 2018 May 31;378(22):2078-2092. doi: 10.1056/NEJMoa1801005. Epub 2018 Apr 16. PMID 29658856
- [Background] Herbst RS, Gordon MS, Fine GD, Sosman JA, Soria JC, Hamid O, et al. A study of MPDL3280A, an engineered PD-L1 antibody in patients with locally advanced or metastatic tumours [abstract 3000]. J Clin Oncol 2013;31(Suppl 15)
- [Background] Hirano F, Kaneko K, Tamura H, Dong H, Wang S, Ichikawa M, Rietz C, Flies DB, Lau JS, Zhu G, Tamada K, Chen L. Blockade of B7-H1 and PD-1 by monoclonal antibodies potentiates cancer therapeutic immunity. Cancer Res. 2005 Feb 1;65(3):1089-96. PMID 15705911
- [Background] Hodi FS, Sznol M, Kluger HM, McDermott DF, Carvajal RD, Lawrence DP et al. Long-term survival of ipilimumab-naive patients (pts) with advanced melanoma (MEL) treated with nivolumab (anti-PD-1, BMS-936558, ONO-4538) in a Phase I trial [ASCO abstract 9002]. J Clin Oncol 2014; 32(Suppl)
- [Background] Iwai Y, Ishida M, Tanaka Y, Okazaki T, Honjo T, Minato N. Involvement of PD-L1 on tumor cells in the escape from host immune system and tumor immunotherapy by PD-L1 blockade. Proc Natl Acad Sci U S A. 2002 Sep 17;99(19):12293-7. doi: 10.1073/pnas.192461099. Epub 2002 Sep 6. PMID 12218188
- [Background] Keir ME, Butte MJ, Freeman GJ, Sharpe AH. PD-1 and its ligands in tolerance and immunity. Annu Rev Immunol. 2008;26:677-704. doi: 10.1146/annurev.immunol.26.021607.090331. PMID 18173375
- [Background] Kong FM, Ritter T, Quint DJ, Senan S, Gaspar LE, Komaki RU, Hurkmans CW, Timmerman R, Bezjak A, Bradley JD, Movsas B, Marsh L, Okunieff P, Choy H, Curran WJ Jr. Consideration of dose limits for organs at risk of thoracic radiotherapy: atlas for lung, proximal bronchial tree, esophagus, spinal cord, ribs, and brachial plexus. Int J Radiat Oncol Biol Phys. 2011 Dec 1;81(5):1442-57. doi: 10.1016/j.ijrobp.2010.07.1977. Epub 2010 Oct 8. PMID 20934273
- [Background] Lan KKG, DeMets DL. Discrete sequential boundaries for clinical trials. Biometrika 1983;70:659-63
- [Background] Lesterhuis WJ, Punt CJ, Hato SV, Eleveld-Trancikova D, Jansen BJ, Nierkens S, Schreibelt G, de Boer A, Van Herpen CM, Kaanders JH, van Krieken JH, Adema GJ, Figdor CG, de Vries IJ. Platinum-based drugs disrupt STAT6-mediated suppression of immune responses against cancer in humans and mice. J Clin Invest. 2011 Aug;121(8):3100-8. doi: 10.1172/JCI43656. Epub 2011 Jul 18. PMID 21765211
- [Background] Lin SH, Lin Y, Price J, Parker M, et al. DETERRED: PD-L1 blockade to evaluate the safety of lung cancer therapy using carboplatin, paclitaxel, and radiation combined with MPDL3280A (atezolizumab). Journal of Clinical Oncology 2017 35:15_suppl, 3064-3064
- [Background] Marks LB, Yorke ED, Jackson A, Ten Haken RK, Constine LS, Eisbruch A, Bentzen SM, Nam J, Deasy JO. Use of normal tissue complication probability models in the clinic. Int J Radiat Oncol Biol Phys. 2010 Mar 1;76(3 Suppl):S10-9. doi: 10.1016/j.ijrobp.2009.07.1754. PMID 20171502
- [Background] Marks LB, Bentzen SM, Deasy JO, Kong FM, Bradley JD, Vogelius IS, El Naqa I, Hubbs JL, Lebesque JV, Timmerman RD, Martel MK, Jackson A. Radiation dose-volume effects in the lung. Int J Radiat Oncol Biol Phys. 2010 Mar 1;76(3 Suppl):S70-6. doi: 10.1016/j.ijrobp.2009.06.091. PMID 20171521
- [Background] Narwal R, Roskos LK, Robbie GJ. Population pharmacokinetics of sifalimumab, an investigational anti-interferon-alpha monoclonal antibody, in systemic lupus erythematosus. Clin Pharmacokinet. 2013 Nov;52(11):1017-27. doi: 10.1007/s40262-013-0085-2. PMID 23754736
- [Background] Nestle U, De Ruysscher D, Ricardi U, Geets X, Belderbos J, Pottgen C, Dziadiuszko R, Peeters S, Lievens Y, Hurkmans C, Slotman B, Ramella S, Faivre-Finn C, McDonald F, Manapov F, Putora PM, LePechoux C, Van Houtte P. ESTRO ACROP guidelines for target volume definition in the treatment of locally advanced non-small cell lung cancer. Radiother Oncol. 2018 Apr;127(1):1-5. doi: 10.1016/j.radonc.2018.02.023. Epub 2018 Mar 28. PMID 29605476
- [Background] Ng CM, Lum BL, Gimenez V, Kelsey S, Allison D. Rationale for fixed dosing of pertuzumab in cancer patients based on population pharmacokinetic analysis. Pharm Res. 2006 Jun;23(6):1275-84. doi: 10.1007/s11095-006-0205-x. Epub 2006 May 26. PMID 16715358
- [Background] Okudaira K, Hokari R, Tsuzuki Y, Okada Y, Komoto S, Watanabe C, Kurihara C, Kawaguchi A, Nagao S, Azuma M, Yagita H, Miura S. Blockade of B7-H1 or B7-DC induces an anti-tumor effect in a mouse pancreatic cancer model. Int J Oncol. 2009 Oct;35(4):741-9. doi: 10.3892/ijo_00000387. PMID 19724910
- [Background] Pardoll DM. The blockade of immune checkpoints in cancer immunotherapy. Nat Rev Cancer. 2012 Mar 22;12(4):252-64. doi: 10.1038/nrc3239. PMID 22437870
- [Background] Paterson AM, Brown KE, Keir ME, Vanguri VK, Riella LV, Chandraker A, Sayegh MH, Blazar BR, Freeman GJ, Sharpe AH. The programmed death-1 ligand 1:B7-1 pathway restrains diabetogenic effector T cells in vivo. J Immunol. 2011 Aug 1;187(3):1097-105. doi: 10.4049/jimmunol.1003496. Epub 2011 Jun 22. PMID 21697456
- [Background] Paz-Ares L, Luft A, Vicente D, Tafreshi A, Gumus M, Mazieres J, Hermes B, Cay Senler F, Csoszi T, Fulop A, Rodriguez-Cid J, Wilson J, Sugawara S, Kato T, Lee KH, Cheng Y, Novello S, Halmos B, Li X, Lubiniecki GM, Piperdi B, Kowalski DM; KEYNOTE-407 Investigators. Pembrolizumab plus Chemotherapy for Squamous Non-Small-Cell Lung Cancer. N Engl J Med. 2018 Nov 22;379(21):2040-2051. doi: 10.1056/NEJMoa1810865. Epub 2018 Sep 25. PMID 30280635
- [Background] Peters S, De Ruysscher D, Dafni U, et al. Safety evaluation of nivolumab added concurrently to radiotherapy in a standard first line chemo-RT regimen in unresectable locally advanced NSCLC: The ETOP NICOLAS phase II trial. J Clin Oncol 36, 2018 (suppl; abstr 8510)
- [Background] Powles T, Eder JP, Fine GD, Braiteh FS, Loriot Y, Cruz C, Bellmunt J, Burris HA, Petrylak DP, Teng SL, Shen X, Boyd Z, Hegde PS, Chen DS, Vogelzang NJ. MPDL3280A (anti-PD-L1) treatment leads to clinical activity in metastatic bladder cancer. Nature. 2014 Nov 27;515(7528):558-62. doi: 10.1038/nature13904. PMID 25428503
- [Background] Rizvi N, Brahmer J, Ou S-H, Segal NH, Khleif SN, Hwu WJ. Safety and clinical activity of MEDI4736, an anti-programmed cell death-ligand-1 (PD-L1) antibody, in patients with nonsmall cell lung cancer (NSCLC). J Clin Oncol 2015;33:Abstract 8032
- [Background] Roselli M, Cereda V, di Bari MG, Formica V, Spila A, Jochems C, Farsaci B, Donahue R, Gulley JL, Schlom J, Guadagni F. Effects of conventional therapeutic interventions on the number and function of regulatory T cells. Oncoimmunology. 2013 Oct 1;2(10):e27025. doi: 10.4161/onci.27025. PMID 24353914
- [Background] Schadendorf D, Hodi FS, Robert C et al. Pooled analysis of long-term survival data from phase II and phase III trials of ipilimumab in metastatic or locally advanced, unresectable melanoma [abstract 24]. Presented at European Cancer Congress 2013 (ECCO-ESMO-ESTRO); 27 September to 01 October 2013; Amsterdam, The Netherlands
- [Background] Segal NH, Ou S-HI, Balmanoukian AS, Fury MG, Massarelli E, Brahmer JR, et al. Safety and efficacy of MEDI4736, an anti-PD-L1 antibody, in patients from a squamous cell carcinoma of the head and neck (SCCHN) expansion cohort. J Clin Oncol 2015;33:Abstract 3011
- [Background] Senan S, Brade A, Wang LH, Vansteenkiste J, Dakhil S, Biesma B, Martinez Aguillo M, Aerts J, Govindan R, Rubio-Viqueira B, Lewanski C, Gandara D, Choy H, Mok T, Hossain A, Iscoe N, Treat J, Koustenis A, San Antonio B, Chouaki N, Vokes E. PROCLAIM: Randomized Phase III Trial of Pemetrexed-Cisplatin or Etoposide-Cisplatin Plus Thoracic Radiation Therapy Followed by Consolidation Chemotherapy in Locally Advanced Nonsquamous Non-Small-Cell Lung Cancer. J Clin Oncol. 2016 Mar 20;34(9):953-62. doi: 10.1200/JCO.2015.64.8824. Epub 2016 Jan 25. PMID 26811519
- [Background] Simon R. Optimal two-stage designs for phase II clinical trials. Control Clin Trials. 1989 Mar;10(1):1-10. doi: 10.1016/0197-2456(89)90015-9. PMID 2702835
- [Background] Socinski MA, Jotte RM, Cappuzzo F, Orlandi F, Stroyakovskiy D, Nogami N, Rodriguez-Abreu D, Moro-Sibilot D, Thomas CA, Barlesi F, Finley G, Kelsch C, Lee A, Coleman S, Deng Y, Shen Y, Kowanetz M, Lopez-Chavez A, Sandler A, Reck M; IMpower150 Study Group. Atezolizumab for First-Line Treatment of Metastatic Nonsquamous NSCLC. N Engl J Med. 2018 Jun 14;378(24):2288-2301. doi: 10.1056/NEJMoa1716948. Epub 2018 Jun 4. PMID 29863955
- [Background] Steuer CE, Behera M, Ernani V, Higgins KA, Saba NF, Shin DM, Pakkala S, Pillai RN, Owonikoko TK, Curran WJ, Belani CP, Khuri FR, Ramalingam SS. Comparison of Concurrent Use of Thoracic Radiation With Either Carboplatin-Paclitaxel or Cisplatin-Etoposide for Patients With Stage III Non-Small-Cell Lung Cancer: A Systematic Review. JAMA Oncol. 2017 Aug 1;3(8):1120-1129. doi: 10.1001/jamaoncol.2016.4280. PMID 27978552
- [Background] Stewart R, Morrow M, Hammond SA, Mulgrew K, Marcus D, Poon E, Watkins A, Mullins S, Chodorge M, Andrews J, Bannister D, Dick E, Crawford N, Parmentier J, Alimzhanov M, Babcook JS, Foltz IN, Buchanan A, Bedian V, Wilkinson RW, McCourt M. Identification and Characterization of MEDI4736, an Antagonistic Anti-PD-L1 Monoclonal Antibody. Cancer Immunol Res. 2015 Sep;3(9):1052-62. doi: 10.1158/2326-6066.CIR-14-0191. Epub 2015 May 5. PMID 25943534
- [Background] Tarhini AA, Kirkwood JM. Tremelimumab (CP-675,206): a fully human anticytotoxic T lymphocyte-associated antigen 4 monoclonal antibody for treatment of patients with advanced cancers. Expert Opin Biol Ther. 2008 Oct;8(10):1583-93. doi: 10.1517/14712598.8.10.1583. PMID 18774925
- [Background] Topalian SL, Hodi FS, Brahmer JR, Gettinger SN, Smith DC, McDermott DF, Powderly JD, Carvajal RD, Sosman JA, Atkins MB, Leming PD, Spigel DR, Antonia SJ, Horn L, Drake CG, Pardoll DM, Chen L, Sharfman WH, Anders RA, Taube JM, McMiller TL, Xu H, Korman AJ, Jure-Kunkel M, Agrawal S, McDonald D, Kollia GD, Gupta A, Wigginton JM, Sznol M. Safety, activity, and immune correlates of anti-PD-1 antibody in cancer. N Engl J Med. 2012 Jun 28;366(26):2443-54. doi: 10.1056/NEJMoa1200690. Epub 2012 Jun 2. PMID 22658127
- [Background] Topalian SL, Sznol M, McDermott DF, Kluger HM, Carvajal RD, Sharfman WH, Brahmer JR, Lawrence DP, Atkins MB, Powderly JD, Leming PD, Lipson EJ, Puzanov I, Smith DC, Taube JM, Wigginton JM, Kollia GD, Gupta A, Pardoll DM, Sosman JA, Hodi FS. Survival, durable tumor remission, and long-term safety in patients with advanced melanoma receiving nivolumab. J Clin Oncol. 2014 Apr 1;32(10):1020-30. doi: 10.1200/JCO.2013.53.0105. Epub 2014 Mar 3. PMID 24590637
- [Background] Tsujino K, Kurata T, Yamamoto S, Kawaguchi T, Kubo A, Isa S, Hasegawa Y, Ou SH, Takada M, Ando M. Is consolidation chemotherapy after concurrent chemo-radiotherapy beneficial for patients with locally advanced non-small-cell lung cancer? A pooled analysis of the literature. J Thorac Oncol. 2013 Sep;8(9):1181-9. doi: 10.1097/JTO.0b013e3182988348. PMID 23883782
- [Background] Wang DD, Zhang S, Zhao H, Men AY, Parivar K. Fixed dosing versus body size-based dosing of monoclonal antibodies in adult clinical trials. J Clin Pharmacol. 2009 Sep;49(9):1012-24. doi: 10.1177/0091270009337512. Epub 2009 Jul 20. PMID 19620385
- [Background] Wang E, Kang D, Bae KS, Marshall MA, Pavlov D, Parivar K. Population pharmacokinetic and pharmacodynamic analysis of tremelimumab in patients with metastatic melanoma. J Clin Pharmacol. 2014 Oct;54(10):1108-16. doi: 10.1002/jcph.309. Epub 2014 Apr 23. PMID 24737343
- [Background] Wang Z, Till B, Gao Q. Chemotherapeutic agent-mediated elimination of myeloid-derived suppressor cells. Oncoimmunology. 2017 Jun 16;6(7):e1331807. doi: 10.1080/2162402X.2017.1331807. eCollection 2017. PMID 28811975
- [Background] Wang K, Eblan MJ, Deal AM, Lipner M, Zagar TM, Wang Y, Mavroidis P, Lee CB, Jensen BC, Rosenman JG, Socinski MA, Stinchcombe TE, Marks LB. Cardiac Toxicity After Radiotherapy for Stage III Non-Small-Cell Lung Cancer: Pooled Analysis of Dose-Escalation Trials Delivering 70 to 90 Gy. J Clin Oncol. 2017 May 1;35(13):1387-1394. doi: 10.1200/JCO.2016.70.0229. Epub 2017 Jan 23. PMID 28113017
- [Background] Wiens BL. A fixed sequence Bonferroni procedure for testing multiple endpoints Pharmaceut. Statist. 2003; 2: 211-215
- [Background] Wolchok JD, Kluger H, Callahan MK, Postow MA, Rizvi NA, Lesokhin AM, Segal NH, Ariyan CE, Gordon RA, Reed K, Burke MM, Caldwell A, Kronenberg SA, Agunwamba BU, Zhang X, Lowy I, Inzunza HD, Feely W, Horak CE, Hong Q, Korman AJ, Wigginton JM, Gupta A, Sznol M. Nivolumab plus ipilimumab in advanced melanoma. N Engl J Med. 2013 Jul 11;369(2):122-33. doi: 10.1056/NEJMoa1302369. Epub 2013 Jun 2. PMID 23724867
- [Background] Yuan J, Adamow M, Ginsberg BA, Rasalan TS, Ritter E, Gallardo HF, Xu Y, Pogoriler E, Terzulli SL, Kuk D, Panageas KS, Ritter G, Sznol M, Halaban R, Jungbluth AA, Allison JP, Old LJ, Wolchok JD, Gnjatic S. Integrated NY-ESO-1 antibody and CD8+ T-cell responses correlate with clinical benefit in advanced melanoma patients treated with ipilimumab. Proc Natl Acad Sci U S A. 2011 Oct 4;108(40):16723-8. doi: 10.1073/pnas.1110814108. Epub 2011 Sep 20. PMID 21933959
- [Background] Zhang C, Wu S, Xue X, Li M, Qin X, Li W, Han W, Zhang Y. Anti-tumor immunotherapy by blockade of the PD-1/PD-L1 pathway with recombinant human PD-1-IgV. Cytotherapy. 2008;10(7):711-9. doi: 10.1080/14653240802320237. PMID 18841514
- [Background] Zhang S, Shi R, Li C, Parivar K, Wang DD. Fixed dosing versus body size-based dosing of therapeutic peptides and proteins in adults. J Clin Pharmacol. 2012 Jan;52(1):18-28. doi: 10.1177/0091270010388648. Epub 2011 Jan 13. PMID 21233304
- [Background] Zou W, Chen L. Inhibitory B7-family molecules in the tumour microenvironment. Nat Rev Immunol. 2008 Jun;8(6):467-77. doi: 10.1038/nri2326. PMID 18500231
- See also: NCCN Guidelines for Treatment of Non-Small Cell Lung Cancer — https://www.nccn.org/store/login/login.aspx?ReturnURL=https://www.nccn.org/professionals/physician_gls/pdf/nscl.pdf